CLINICAL TRIAL: NCT01832805
Title: The Effects of Thetaburst Stimulation in Treatment Resistant Unipolar Depressed Patients
Brief Title: Theta Burst Study Ghent
Acronym: TBS Ghent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013/392
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Unipolar Major Depression
Keywords: depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Theta burst stimulation (Experimental): Specific developed sham coil.
  Interventions: Other: Theta burst stimulation.

INTERVENTIONS:
Other: Theta burst stimulation. — In each session, subjects will receive 54 Theta burst trains of 2 seconds duration, separated by an intertrain interval of 18 seconds, delivered on the left dorsolateral prefrontal cortex (DLPFC). The treatment protocol of in total 20 Theta burst sessions will be spread over 4 days, yielding a total of 32400 stimuli. On each stimulation day, a given patient shall receive 5 sessions with a between session delay of 10 to 15 minutes.

SUMMARY:
50 Right-handed antidepressant-free unipolar depressed patients (age 18-65 years) will be treated with in total 20 Theta burst sessions; these will be spread over 4 days. On each stimulation day, a given patient shall receive 5 sessions with a between session delay of 10 to 15 minutes. Patients will be selected using the structured Mini-International Neuropsychiatric Interview (MINI). All will be at least stage I treatment resistant. Because concomitant antidepressant treatment can confound outcome results, all patients will go through a medication washout before entering the study and they will be free from any antidepressant, neuroleptic and mood stabilizer for at least two weeks before entering the treatment protocol. Only habitual benzodiazepine agents will be allowed.

All patients will be closely matched for gender and age with 50 never-depressed medication-free healthy volunteers. Only baseline measurements will be collected: no volunteer will undergo the treatment.

We expect that real Theta burst treatment and not sham will result in a significant and clinical meaningful response.

ELIGIBILITY:
Inclusion Criteria:

* antidepressant-free unipolar depression
* age between 18 and 65 years
* right handed
* at least stage I treatment resistant

Exclusion Criteria:

* current or past history of epilepsy, neurosurgical interventions, having a pacemaker or metal or magnetic objects in the brain, alcohol dependence and suicide attempts within 6 months before the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Depression severity in Theta burst treatment at baseline. | At baseline.
  Depression severity will be assessed, using the 21-item Beck Depression Inventory (BDI-II) and the 17-item Hamilton Depression Rating Scale (HDRS).
Depression severity of Theta burst treatment after 1 week of treatment. | After 1 week of TBS-rTMS/sham treatment.
  Depression severity will be assessed, using the 21-item Beck Depression Inventory (BDI-II) and the 17-item Hamilton Depression Rating Scale (HDRS).
Depression severity will be assessed at the end of the final second week of the stimulation protocol. | At the end of the final second week of the stimulation protocol.
  Depression severity will be assessed, using the 21-item Beck Depression Inventory (BDI-II) and the 17-item Hamilton Depression Rating Scale (HDRS).
Depression severity will be assessed two weeks after stimulation. | Two weeks after stimulation.
  Depression severity will be assessed, using the 21-item Beck Depression Inventory (BDI-II) and the 17-item Hamilton Depression Rating Scale (HDRS).
Suicidal ideation will be assessed at baseline. | At baseline.
  Suicidal ideation will be assessed with the suicidal ideation scale (SSI).
Suicidal ideation will be assessed after 1 week of treatment. | After 1 week of TBS-rTMS/sham treatment.
  Suicidal ideation will be assessed using the suicidal ideation scale (SSI).
Suicidal ideation will be assessed at the end of the final second week of the stimulation protocol. | At the end of the final second week of the stimulation protocol.
  Suicidal ideation will be assessed using the suicidal ideation scale (SSI).
Suicidal ideation will be assessed two weeks after stimulation. | Two weeks after stimulation.
  Suicidal ideation will be assessed using the suicidal ideation scale (SSI).

SECONDARY OUTCOMES:
Resting state functional connectivity; diffusion MRI at baseline. | At baseline.
  Siemens 3T MRI.
Resting state functional connectivity; diffusion MRI after 1 week of treatment. | After 1 week of TBS-rTMS/sham treatment.
  Siemens 3T MRI.
Resting state functional connectivity; diffusion MRI at the end of the final second week of the stimulation protocol. | At the end of the final second week of the stimulation protocol.
  Siemens 3T MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Desmyter, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Wu GR, Duprat R, Baeken C. Accelerated iTBS changes perfusion patterns in medication resistant depression. J Affect Disord. 2022 Jun 1;306:276-280. doi: 10.1016/j.jad.2022.03.036. Epub 2022 Mar 16. PMID 35306123
- [Derived] Wu GR, Baeken C. Individual interregional perfusion between the left dorsolateral prefrontal cortex stimulation targets and the subgenual anterior cortex predicts response and remission to aiTBS treatment in medication-resistant depression: The influence of behavioral inhibition. Brain Stimul. 2022 Jan-Feb;15(1):182-189. doi: 10.1016/j.brs.2021.12.003. Epub 2021 Dec 10. PMID 34902623
- [Derived] Baeken C, van Beek V, Vanderhasselt MA, Duprat R, Klooster D. Cortical Thickness in the Right Anterior Cingulate Cortex Relates to Clinical Response to Left Prefrontal Accelerated Intermittent Theta Burst Stimulation: An Exploratory Study. Neuromodulation. 2021 Jul;24(5):938-949. doi: 10.1111/ner.13380. Epub 2021 Mar 31. PMID 33788975
- [Derived] Baeken C, Wu G, Sackeim HA. Accelerated iTBS treatment applied to the left DLPFC in depressed patients results in a rapid volume increase in the left hippocampal dentate gyrus, not driven by brain perfusion. Brain Stimul. 2020 Sep-Oct;13(5):1211-1217. doi: 10.1016/j.brs.2020.05.015. Epub 2020 Jun 5. PMID 32512184
- [Derived] Klooster DC, Vos IN, Caeyenberghs K, Leemans A, David S, Besseling RM, Aldenkamp AP, Baeken C. Indirect frontocingulate structural connectivity predicts clinical response to accelerated rTMS in major depressive disorder. J Psychiatry Neurosci. 2020 Jul 1;45(4):243-252. doi: 10.1503/jpn.190088. PMID 31990490
- [Derived] Wu GR, Wang X, Baeken C. Baseline functional connectivity may predict placebo responses to accelerated rTMS treatment in major depression. Hum Brain Mapp. 2020 Feb 15;41(3):632-639. doi: 10.1002/hbm.24828. Epub 2019 Oct 21. PMID 31633261
- [Derived] Baeken C, Wu GR, van Heeringen K. Placebo aiTBS attenuates suicidal ideation and frontopolar cortical perfusion in major depression. Transl Psychiatry. 2019 Jan 29;9(1):38. doi: 10.1038/s41398-019-0377-x. PMID 30696807
- [Derived] Baeken C, Duprat R, Wu GR, De Raedt R, van Heeringen K. Subgenual Anterior Cingulate-Medial Orbitofrontal Functional Connectivity in Medication-Resistant Major Depression: A Neurobiological Marker for Accelerated Intermittent Theta Burst Stimulation Treatment? Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Oct;2(7):556-565. doi: 10.1016/j.bpsc.2017.01.001. Epub 2017 Jan 20. PMID 29560909
- [Derived] Desmyter S, Duprat R, Baeken C, Van Autreve S, Audenaert K, van Heeringen K. Accelerated Intermittent Theta Burst Stimulation for Suicide Risk in Therapy-Resistant Depressed Patients: A Randomized, Sham-Controlled Trial. Front Hum Neurosci. 2016 Sep 27;10:480. doi: 10.3389/fnhum.2016.00480. eCollection 2016. PMID 27729854
- See also: Related Info — http://www.uzgent.be